CLINICAL TRIAL: NCT05078853
Title: Thyroglobulin Point of Care Assay for Rapid Detection of Metastatic Differentiated Thyroid Carcinoma- A Multi-Center Validation Study
Brief Title: Thyroglobulin Point of Care Assay for Rapid Detection of Metastatic Differentiated Thyroid Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Uri Yoel MD, Dr.Uri Yoel, Soroka University Medical Center
Other Study IDs: SCRC21021CTIL
Record Dates: First submitted 2021-09-27; First posted 2021-10-15 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Differentiated Thyroid Cancer; Lymph Node Metastases
Keywords: Differentiated thyroid carcinoma; Papillary thyroid carcinoma; Cervical lymph nodes metastases; Thyroglobulin washout; Point of care assay
MeSH Terms: conditions — Lymphatic Metastasis; Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — FNA washout from cervical lymph node suspected as differentiated thyroid carcinoma metastasis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Formal/standard evaluation of a suspected cervical lymph node: Patient with cervical lymph node suspected as differentiated thyroid carcinoma metastasis will be evaluated according to the current accepted American Thyroid Association Guidelines.
  Two clinical scenarios, for each one of them the formal evaluation is described below:
  1. Fine needle aspiration Clinic (a patient with known or suspected differentiated thyroid carcinoma is evaluation for suspicious cervical lymph node): the formal evaluation will include cytology and formal thyroglobulin measurement from the needle washout.
  2. Operating room (evaluation of suspicious cervical lymph node found during partial or complete thyroidectomy in patient with known or suspected differentiated thyroid carcinoma): the formal evaluation will include frozen section and/or final histology.
- Point of care assay for thyroglobulin (POC-Tg) evaluation of a suspected cervical lymph node: Patient with cervical lymph node suspected as differentiated thyroid carcinoma metastasis will be evaluated using the study kit: Novel rapid POC-Tg.
  Two clinical scenarios, for each one of them the performance of the study kit (POC-Tg) will be valuated in parallel to the formal evaluation:
  1. Fine needle aspiration Clinic (a patient with known or suspected differentiated thyroid carcinoma is evaluation for suspicious cervical lymph node): the suspected cervical lymph node will be evaluated using the POC-Tg in parallel to the formal evaluation.
  2. Operating room (evaluation of suspicious cervical lymph node found during partial or complete thyroidectomy in patient with known or suspected differentiated thyroid carcinoma): the suspected cervical lymph node will be evaluated using the POC-Tg in parallel to the formal evaluation.
  Interventions: Device: Point of care assay for thyroglobulin (POC-Tg) evaluation of a suspected cervical lymph node

INTERVENTIONS:
Device: Point of care assay for thyroglobulin (POC-Tg) evaluation of a suspected cervical lymph node — FNA Clinic: When a bloody material is seen in the needle, 100 µL of 0.9% saline is drawn via the needle into the syringe. The aspirate is then transferred into an Eppendorf tube. 40 µL is aspirated from the Eppendorf tube and dripped into the middle of the sample well of the POC-Tg kit. Two drops of the buffer are then dispensed into the middle of the sample well. The result of the POC-Tg is obtained and documented after 10 minutes. To compare the accuracy of the POC-Tg kit to the formal immunoassay for Tg, 0.9% saline is added to the aspirate that was left in the Eppendorf tube to a final volume of 0.6 mL. This volume is transferred into a gel containing tube and sent to the clinical laboratory that performs Tg measurement.
  Operating room: When an indeterminate or suspicious LN is found, the LN is dissected and evaluated by both the formal evaluation and the POC-Tg. Following dissection of the LN, the ex-vivo POC-Tg is conducted as described above.
  Other Names: POC-Tg
  Groups: Point of care assay for thyroglobulin (POC-Tg) evaluation of a suspected cervical lymph node

SUMMARY:
Background: Despite a favorable prognosis, metastatic cervical lymph nodes (LN), are not uncommon among patients with differentiated thyroid cancer (DTC). Current guidelines recommend that a suspicious cervical LN on neck ultrasound (US) should be investigated with fine needle aspiration biopsy for cytology (FNAC) and for thyroglobulin (Tg) measurement (FNA-Tg), using saline washout of the needle content. Since Tg is a protein produced exclusively by thyroid follicular cells, a positive FNA-Tg result establishes the diagnosis of metastatic DTC. Currently, following LN biopsy, a patient must wait days to weeks to receive results, that directly impacts the treatment plan. This delay may be solved by a point of care assay of the washout Tg (POC-Tg), drawn from a suspicious cervical LN. Another potential novel usage of POC-Tg is the evaluation of suspicious LN found during neck surgery for known or suspicious DTC. Here, the POC-Tg may save the time needed for the completion of 'frozen section'.

The study product: POC-Tg is a lateral flow immunoassay for Tg, able to detect within minutes Tg at concentration equal to 5 ng/mL and above (the midrange of the accepted cut-off).

Methods: The multi-center validation study will include 100 patients in the FNA clinic, and 150 LN (dissected from 50-150 patients) in the operating room (OR). Each LN will be evaluated using both the formal accepted method (in the FNA clinic, the combination of FNAC and FNA-Tg; and frozen section in the OR), and the novel POC-Tg. Clinical decisions will be made according to the formal evaluation only. In a retrospective analysis, the investigators will estimate the sensitivity and specificity of the POC-Tg and the formal accepted method against the reference ('gold') standard (cytology, histology and follow-up US in the FNA clinic setting, and final histology in the OR setting).

DETAILED DESCRIPTION:
Methods and materials

Hypothesis: The diagnostic accuracy of the novel POC-Tg will be comparable with the current diagnostic methods used for the evaluation of cervical LNs suspected as DTC metastases.

Aim

1. To validate the POC-Tg in the FNA clinic: Indeterminate or suspicious cervical LNs in patients with known or suspected DTC will be assessed using both the novel POC-Tg, and the formal evaluation (formal immunoassay for Tg and cytology).
2. To validate the POC-Tg in the OR: Indeterminate or suspicious cervical LNs in patients operated for DTC will be assessed using both the novel POC-Tg and the formal evaluation (frozen section and/or final histology in the pathological institution).

Significance: An accurate POC-Tg may change current diagnostic and treatment approaches of patients with suspected metastatic DTC and improve patient management.

Study design:

The investigators will conduct a multi-center study. All coded data will be managed centrally, using an electronic case report form, by Soroka University Medical Center (SUMC) Clinical Research Center. All the data for sensitivity and specificity evaluations of the novel POC-Tg, and the current diagnostic methods of DTC cervical LN metastasis will be analyzed retrospectively against the reference ('gold') standard (see below). Clinical decisions will be made according to the current guidelines and accepted approaches for the evaluation of cervical LN that are suspected as DTC metastases (in the FNA clinic, the combination of FNAC and FNA-Tg; and in the OR, frozen section and/or final histology).

Detailed Study Protocol

1. The FNA clinic arm:

   All recruited patients will undergo US examination of the neck using an US scanner with a 12.5-MHz linear phased-array transducer. US-guided FNA of suspicious or indeterminate LN will be performed by an experienced physician (an endocrinologist, otolaryngologist, or a radiologist), as clinically indicated. LN will be classified as suspicious if any of the following imaging features is present: calcification, cystic change, hyper-echogenicity, or peripheral or diffuse increased vascularity on color Doppler imaging. LN will be classified as indeterminate suspicious when neither clear benign nor suspicious imaging features are found (neither echogenic hilum nor hilar vascularity in the absence of suspicious findings). The FNA procedure will be performed under US guidance with the free hand technique using a 22 to 25-gauge needle connected to a 3 to 10-mL syringe, as routinely performed in each medical center. If technically and clinically possible, each LN will be sampled twice: one passage for cytology and one passage for FNA-Tg washout.

   FNA for cytology (FNAC)- FNAC specimens will be prepared from direct smears and/or liquid-based cytology, as routinely performed in each medical center. In the FNA clinic at SUMC, specimens will be smeared on slides and immediately fixed in 95% ethanol using the direct smear method. With the liquid-based cytology method, specimens will be prepared using the ThinPrep PreservCyt® (Hologic Ins., Marlborough, MA, USA). Cytology findings will be interpreted by cytopathologists specialized in thyroid cytology. The cytology results obtained from the LN of interest will be categorized as: malignant, benign, or indeterminate.

   FNA-Tg and POC-Tg- After the needle is localized inside the LN of interest, a negative pressure will be produced by the syringe handle, while performing inward-outward and rotatory movement, until a bloody material is seen in the proximal end of the needle. Thereafter, 100 µL of 0.9% (w/v) saline will be drawn via the needle into the syringe that will contain 100 µL of mildly bloody aspirate from the LN of interest. The aspirate will then be transferred into an Eppendorf tube through the same needle that was used for the FNA procedure. At this time the product bag of the POC-Tg kit will be opened. Using a disposable pipette, 40 µL will be aspirated from the Eppendorf tube and dripped into the middle of the sample well of the POC-Tg kit. Two drops of the buffer will then be dispensed into the middle of the sample well. Results of the POC-Tg will be obtained and documented after 10 minutes. To compare the accuracy of the POC-Tg kit to the formal immunoassay for Tg that is used in each institution, 0.9% saline will be added to the aspirate that will be left in the Eppendorf tube to a final volume of 0.6 mL, then transferred into a gel containing tube and sent to the clinical laboratory that performs Tg measurement.

   Reference ('gold') Standard- LN will be finally diagnosed as metastatic if they show malignant FNA cytology (Bethesda 6) or meeting at least one of the following criteria: (i) malignancy confirmation based on the surgical specimen (histology), (ii) subsequent repeat FNA or core-needle biopsy reporting Bethesda 6 or DTC, respectively, or (iii) follow-up with imaging after one year showing clear US features of metastasis. LN with benign or indeterminate FNA cytology free of metastatic disease by the same criteria will be finally diagnosed as benign.

   Routine laboratory assessment- Analytes as plasma Tg, anti-Tg-antibodies, anti-thyroid-peroxidase, TSH, free T4, and free T3 will be performed as part of the routine evaluation of patients with suspected or known thyroid disease.

   Required data (data to capture):
   * Technical data (per center): The firm of the US used in each institution, type of FNA-Tg immunoassay (type, firm, limit of detection, reported accuracy), cytological evaluation used (type and firm).
   * Demographic and clinical data: Date of birth, date of the index procedure, age (years) at the time of the index procedure, past diagnosis of Hashimoto thyroiditis (ICD9 code 2452), past diagnosis of Grave's disease (ICD9 code 2420), treated with levothyroxine or an anti-thyroid-drug, prior thyroid surgery (no, lobectomy [left/right], sub-total thyroidectomy, complete thyroidectomy), prior neck dissection (central [no, right, left], lateral level 2-4 [no, right, left], lateral level 5 [no, right, left]).
   * Laboratory data prior to the index procedure (each will be reported with units used by the laboratory where it was performed, and as X upper limit of norm): TSH, Tg, anti-Tg- antibodies, free T4, free T3, anti-thyroid peroxidase.
   * Regarding US findings of the thyroid gland, the following information will be accessed for the most suspicious nodule: TIRADS points, TIRADS class, American Thyroid Association class, three dimensions, and volume.
   * US findings of the LN from which the procedure is done (yes/no for each): echogenic hilum, hilar vascularity, calcification, cystic change, hyper-echogenicity, peripheral or diffuse increased vascularity on color Doppler imaging, final interpretation (indeterminate/suspicious).
   * Cytological report of the most suspicious/relevant thyroid nodule: Bethesda system score.
   * Cytological findings of the LN from which the procedure is done: classified as benign, indeterminate, or malignant.
   * FNA-Tg- units as reported by the institutional lab, and X upper limit of norm.
   * POC-Tg- positive or negative.
   * Final histology
2. The OR arm:

Thyroid/neck surgery and Ex-vivo FNA- All recruited patients will be operated, as clinically indicated, either as part of primary treatment for DTC or for persistent or recurrent DTC. Thyroid and neck dissection surgeries will be led by experienced otolaryngologist or endocrine surgeons. Whenever an indeterminate or suspicious LN is found, and it is deemed that a frozen section report of the LN may change surgery extent, the LN will be dissected and evaluated by both the formal evaluation-frozen section and POC-Tg. Following dissection of the LN, the ex-vivo FNA-Tg and POC-Tg will be conducted as detailed above (under the 'FNA-Tg and POC-Tg' section).

Frozen section- The relevant specimen for frozen section will be dissected, treated, and sent to pathological evaluation as clinically indicated and routinely performed in each medical center. All clinical decisions during the surgery will be made according to the frozen section results or clinical judgment. The histology results of the frozen section analysis, obtained from the LN of interest, will be categorized as: malignant, benign, or indeterminate/inconclusive.

Reference ('gold') Standard- LN will be finally diagnosed as benign or malignant (DTC metastasis) according to the final histological report.

Required data:

* Technical data (per center): Frozen section equipment, type of FNA-Tg immunoassay (type, firm, limit of detection, reported accuracy).
* Demographic and clinical data: Date of birth, date of the index procedure, age (years) at the time of the index procedure, past diagnosis of Hashimoto thyroiditis (ICD9 code 2452), past diagnosis of Grave's disease (ICD9 code 2420), treated with levothyroxine or an anti-thyroid-drug, prior thyroid surgery (no, lobectomy [left/right], sub-total thyroidectomy, complete thyroidectomy), prior neck dissection (central [no, right, left], lateral level 2-4 [no, right, left], lateral level 5 [no, right, left]).
* Laboratory data prior to the index procedure (each will be reported with units used by the laboratory where it was performed, and as X upper limit of norm): TSH, Tg, anti-Tg- antibodies, free T4, free T3, anti-thyroid peroxidase.
* Cytological report of the most suspicious/relevant thyroid nodule: Bethesda system.
* Cytological findings of the relevant LN: classified as benign, indeterminate, or malignant.
* The planned operation: lobectomy [left/right], sub-total thyroidectomy, complete thyroidectomy, neck dissection (central [no, right, left], lateral level 2-4 [no, right, left], lateral level 5[no, right, left]).
* FNA-Tg- units as reported by the institutional lab, and X upper limit of norm.
* POC-Tg- positive or negative.
* The frozen section report: malignant, benign, or indeterminate/inconclusive.
* Overall time needed for the frozen section evaluation - from dissection to report (minutes).
* The operation that was executed: as planned/ extended (specify).
* Final histology

Statistical analysis:

The estimates of sensitivity and specificity will be calculated for the positive and negative samples, respectively, while their status will be defined using the reference ('gold') standard (diagnostic procedure depending on cytology and histology results, and other clinical information). To address the main objectives of the study, the 95% confidence interval will be constructed around each of the validation parameters. A design effect will be considered for the samples taken in the OR that originate from the same patient, using a sandwich estimator of the standard error. Furthermore, the researchers will explore potential factors associated with agreement and disagreement of the diagnostic test with the reference ('gold') standard. Specifically, characteristics of patients in whom the diagnosis was aligned with the reference ('gold') standard will be compared to those with discordant results. This type of analysis will indicate populations, if any, for which the test should not be utilized. The comparisons will be conducted using standard statistical methodology, i.e. Chi-Square or Fisher's Exact test for categorical variables and t-test, ANOVA or non-parametric alternative tests for continuous parameters. Confidence intervals will be adjusted to clustered observations as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are able and agree to sign the informed consent document.
2. Aged 18 years or older.

   In the FNA clinic arm:
3. Patients evaluated for thyroid nodule/s suspected or known as DTC, accompanied by cervical LN/s suspected as DTC metastasis.
4. Patients following treatment for DTC (partial or total thyroidectomy, with or without compartmental neck dissection), with cervical LN/s suspected as DTC recurrency.

   In the OR arm:
5. Patients operated for known DTC (partial or total thyroidectomy, with or without compartmental neck dissection).
6. Patients operated for DTC recurrency ('completion' and/or compartmental neck dissection).

   -

   Exclusion Criteria:

   Pregnant women

   -

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: FNA Clinic: Patients evaluated in FNA clinic for cervical lymph node/s suspected as DTC metastasis.
  Operating room: Patients operated for known or suspected DTC with cervical lymph node/s metastasis.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Accurate diagnosis of cervical lymph node in the FNA clinic being benign or malignant | Up to 1 year following POC-Tg assessment
  Sensitivity and specificity of the POC-Tg for the detection of DTC metastases to cervical LN compared to the current accepted evaluation
Accurate diagnosis of suspicious cervical lymph node in the operating room being benign or malignant | Up to 1 year following POC-Tg assessment
  Sensitivity and specificity of the POC-Tg for the detection of DTC metastases to cervical LN compared to the current accepted evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Uri Yoel, M.D., Principal Investigator — Soroka University Medical Center, Beer Sheva, Israel
Locations (5):
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Soroka University Medical Center, Beersheba
  - Hebrew University Medical Center, Mount Scopus, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - A.R.M Medical Center, Assuta Ramat Hahayal, Tel Aviv